CLINICAL TRIAL: NCT06692816
Title: Clinical Efficacy of Pulsed Electromagnetic Field Therapy (PEMT) in Patients With Degenerative Meniscus Lesions: Double-Blind Randomized Sham-Controlled Study
Brief Title: Pulsed Electromagnetic Field Therapy (PEMT) in Patients With Degenerative Meniscus Lesions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Sevda Adar, Assistant Professor, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAPEMT
Record Dates: First submitted 2024-11-12; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Meniscus Lesion; Pain
MeSH Terms: conditions — Pain | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEMT (Experimental): It was planned for this group to apply PEMT to the painful knee region with an electromagnetic field device (ASA Pmt Quatro Pro, ASA Srl Via A.Volta 9-36057, May, 2012 Arcugnano (VI)-Italia) with a physiotherapist who is trained in using the device and has at least 5 years of experience, at a frequency of 50 Hz, an intensity of 85 Gauss (8.5 milliTesla) and for 30 minutes. The treatment period was planned as a total of 20 sessions, 5 days a week for 4 weeks. As a therapeutic exercise program, it was planned to apply joint range of motion, walking, balance, coordination, cycling, isometric and isotonic strengthening exercises by a trained physiotherapist with at least 5 years of experience and that the patients would do these exercises three times a day, in 3 sets, with 10 repetitions.
  Interventions: Other: Rehabilitation
- SHAM (Sham Comparator): It was planned for this group to receive sham PEMT, with the electromagnetic field device turned off, for a total of 20 sessions, 5 days a week for 4 weeks, for 30 minutes each session, and a therapeutic exercise program, for a total of 20 sessions, 5 days a week for 4 weeks, for 30 minutes each session, including range of motion, walking, balance, coordination, cycling, isometric and isotonic strengthening exercises, by a trained physiotherapist with at least 5 years of experience, and for the patients to do these exercises three times a day, in 3 sets, with 10 repetitions.
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — As a therapeutic exercise program, it was planned to apply joint range of motion, walking, balance, coordination, cycling, isometric and isotonic strengthening exercises by a trained physiotherapist with at least 5 years of experience and that the patients would do these exercises three times a day, in 3 sets, with 10 repetitions.

SUMMARY:
Pulse Electromagnetic Field Therapy (PEMT) is effective in the treatment of many diseases, especially musculoskeletal system diseases, due to its analgesic effect with the effect of induced currents, and also its anti-inflammatory , edema reducing, antispasmodic and blood flow accelerating effects with additional mechanisms. The aim of our study is to evaluate the effects of Pulsed Electromagnetic Field Therapy (PEMT) degenerative To investigate the effects on pain, quality of life and function in patients with meniscal lesions.

DETAILED DESCRIPTION:
Menisci are responsible for carrying the load in the knee joint, transmitting the load, absorbing impacts, lubricating the joint and stabilizing the joint .The menisci to perform their functions properly, the integrity of their anterior and posterior roots at their attachment points on the tibial plateau must be preserved. The male/female ratio of meniscus injuries is 2.5/1, with an incidence of around 60-70 per 100,000. Medial meniscus tears, lateral It is detected 3 times more frequently than meniscus tears. In patients under the age of 30, trauma and in patients over the age of 30, degenerative causes often cause tears.

Meniscus tears can be divided into two groups: traumatic and degenerative . Traumatic tears occur in healthy menisci , most often in young people, as a result of excessive and inappropriate loading. Degenerative tears are common in the elderly, occurring in degenerated menisci under normal load or after minimal trauma . Traumatic injuries most often occur when the body rotates on the knee while the foot is fixed on the ground.

meniscus tears can be divided into two groups : conservative (pharmacological and non -pharmacological) and surgical. Non -pharmacological treatment approaches consist of programs such as patient education, use of assistive devices, lifestyle changes, weight control, and conventional physical therapy methods.

Magnetic Field Therapy is a cheap, non-invasive and safe physical therapy method with no known significant side effects. It is suggested that Pulse Electromagnetic Field Therapy (PEMT) is effective in the treatment of many diseases, especially musculoskeletal system diseases, due to its analgesic effect with the effect of induced currents, and also its anti-inflammatory , edema reducing, antispasmodic and blood flow accelerating effects with additional mechanisms. Current literature suggests that magnetic field therapy may be effective in the treatment of fracture union, knee osteoarthritis , cervical fusion, lumbar and cervical There are studies on its effectiveness in the treatment of various musculoskeletal problems such as discopathy. Pulsed electromagnetic field therapy (PEMT) has been shown to enhance healing of meniscal tears and reduce post- traumatic osteoarthritis in a rat model . However, in the literature Pulsed electromagnetic field therapy (PEMT) degenerative No clinical studies have been found on the effectiveness of meniscus lesions.The aim of our study is to evaluate the effects of Pulsed Electromagnetic Field Therapy (PEMT) degenerative To investigate the effects on pain, quality of life and function in patients with meniscal lesions.

ELIGIBILITY:
Inclusion Criteria:

* Knee pain for at least 2 months
* MRI findings of meniscus degeneration
* The health condition is suitable for rehabilitation
* Ability to understand commands

Exclusion Criteria:

* Inability to cooperate fully and lack of literacy skills
* NSAID use
* Planning pregnancy during pregnancy or treatment process
* A history of physical therapy and rehabilitation for the knee area in the last 6 months.
* A history of local injection treatment to the knee area within the last 6 months,
* A history of trauma, surgery, or fracture in the lower extremity on the side of pain in the last 6 months,
* Lumbar radiculopathy
* Presence of advanced gonarthrosis (Kellgren Lawrence stage 3-4)
* Ligament injury or tear of the knee
* Systemic inflammatory rheumatic disease (rheumatoid arthritis, systemic lupus erythematosus, ankylosing spondylitis, psoriatic arthritis, vasculitis etc.
* Neurological diseases (multiple sclerosis, history of cerebrovascular disease, myopathic diseases, epilepsy, febrile convulsions, etc.),
* Cardiac pacemaker,
* Malignancy,
* Bleeding diathesis,
* An electronic or battery system body implant.
* Acute infections, presence of tuberculosis

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Visual Pain Scale (VAS) - night - rest - movement | Before treatment (T0) At the end of treatment (4 weeks) (T1) At 6 months (T2)
  In treatments applied for knee pain, the primary goal is to focus on the restoration of pain and movement function. Visual Pain Scale (VAS), which is easy to understand, apply and interpret, and provides valid and reliable data in a short time, is the most commonly used method in clinics. With a 100 mm visual linear scale, the patient is told that there is no pain at 0, and that the most severe pain ever felt at 100, and the patient is asked to mark the point corresponding to rest, movement and night pain.
KOOS ( KNEE INJURY AND OSTEOARTHRITIS OUTCOME SCORE) | Before treatment (T0) At the end of treatment (4 weeks) (T1) At 6 months (T2)
  It is a scale used to evaluate symptoms and functional status related to knee injuries and knee osteoarthritis . It has 5 subgroups: pain, daily living activities (ADL), functional status in sports and leisure activities and quality of life related to the knee. Each question is scored with a total of 5 options between 0-4. The average score in each section is multiplied by 100, divided by 4 and subtracted from 100. The possible score varies between 0 and 100 points in each case. A score of 100 indicates no restrictions due to the affected knee , while a score of 0 indicates excessive problems and restrictions.
Lysholm Knee Scoring Scale | Before treatment (T0) At the end of treatment (4 weeks) (T1) At 6 months (T2)
  8 items are asked about symptoms and a total score (0-100) is calculated. A score of 0 indicates the lowest knee function, while a score of 100 indicates the highest knee function. There is a Turkish validity and reliability study.
Western Ontario Meniscus Assessment Questionnaire | Before treatment (T0) At the end of treatment (4 weeks) (T1) At 6 months (T2)
  Physical symptoms experienced by patients due to knee problems are questioned. A total of 16 questions in 3 sections are given 0-10 points. The score for each subgroup is obtained by dividing the marked values of the questions in that section by the number of questions and multiplying by 10. For the total score, all marked values are added, divided by 16 and multiplied by 10. The score is between 0-100. 0 indicates the best symptoms and function, while 100 indicates the worst symptoms and function. There is a Turkish validity and reliability study.

SECONDARY OUTCOMES:
Knee joint range of motion (ROM) | Before treatment (T0) At the end of treatment (4 weeks) (T1) At 6 months (T2)
  In measuring knee range of motion, flexion and extension movements are measured with a goniometer while the patient lies on his back, including active and passive measurements of the knee.
Tegner Activity Level Scale | Before treatment (T0) At the end of treatment (4 weeks) (T1) At 6 months (T2)
  This scale aims to evaluate the activity level of people with knee injuries. The patient's activity is scored between 0 and 10. 0 indicates the lowest activity level, while 10 indicates the highest activity level. There is a Turkish validity and reliability study.
Lower Extremity Y Dynamic Balance Test: | Before treatment (T0) At the end of treatment (4 weeks) (T1) At 6 months (T2)
  Balance is maintained on the Y dynamic balance test platform by keeping the hands fixed on the waist area and the foot fixed at the center point. Then, while maintaining the fixed stance with one foot, the blocks are pushed with the toe tip with the other foot in the anterior (0°), posteromedial (45°) and posterolateral (45°) directions (each time bringing the foot back to the fixed stance point without touching the ground) . After the test is repeated 3 times in each of the three directions ( anterior , posteromedial , posterolateral ), the normalization formula is used. The sum of the 3 directions is divided by 3 times the leg length and multiplied by 100.
SF -36 | Before treatment (T0) At the end of treatment (4 weeks) (T1) At 6 months (T2)
  SF -36 is a generic quality of life scale. It provides the opportunity to ev.aluate the health status of the person in 10 sub-parameters such as physical function, body pain, limitation due to physical problems, emotional well-being, social function, energy/fatigue, general health perception. It contains a total of 36 items. It is evaluated between 0-100 points. It was created to evaluate the health status.
Isokinetic Evaluation of Knee | Before treatment (T0) At the end of treatment (4 weeks) (T1) At 6 months (T2)
  Isokinetic systems are complex systems used for both rehabilitation and patient evaluation. Isokinetic contraction is defined as a contraction at a constant speed throughout the entire range of motion and is equal in speed at every angle of motion. No matter how much force the person applies to the device, they can never exceed the predetermined speed (e.g. 90 degrees per second). The ability to evaluate the desired muscle or muscle groups in isolation and the repeatability and comparability of the measurements are advantageous features.

CONTACTS AND LOCATIONS:
Overall Officials: SEVDA ADAR, Principal Investigator — Afyonkarahisar Health Sciences University

IPD SHARING:
Plan to Share IPD: No